CLINICAL TRIAL: NCT06451757
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Parallel-group, Pivotal Trial to Assess the Efficacy and Safety of Sonlicromanol in Adult Subjects With a Genetically Confirmed Mitochondrial DNA tRNALeu(UUR) m.3243A>G Variant
Brief Title: KHENERFIN Study: A Trial to Evaluate the Efficacy and Safety of Sonlicromanol in Primary Mitochondrial Diseases
Acronym: KH176-301
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Khondrion BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Khondrion B.V.
Expanded Access: Available
Record Dates: First submitted 2024-05-29; First posted 2024-06-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Mitochondrial Diseases; Maternally Inherited Diabetes and Deafness (MIDD); Mitochondrial Encephalomyopathy, Lactic Acidosis and Stroke-like Episodes (MELAS); Mitochondrial DNA tRNALeu(UUR) m.3243A<G Mutation
Keywords: Mitochondrial Diseases; Oxidative Phosphorylation (OXPHOS); Maternally Inherited Diabetes and Deafness (MIDD); Mitochondrial DNA tRNALeu(UUR) m.3243A<G Mutation; Mitochondrial Encephalomyopathy, Lactic Acidosis and Stroke-like episodes (MELAS); Sonlicromanol
MeSH Terms: conditions — Mitochondrial Diseases; Noninsulin-dependent diabetes mellitus with deafness; MELAS Syndrome

STUDY DESIGN:
Intervention Model Description: The study will be a double-blind, randomised, placebo-controlled, multi-centre, parallel-group study. 220 subjects, with a confirmed mitochondrial DNA tRNALeu(UUR) 3243A>G mutation will be randomised in a 1:1 ratio to receive oral administration of 90 mg sonlicromanol (100 mg sonlicromanol.HCl) or placebo twice daily.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial personnel and subjects will be blinded to treatment until the database is locked. Investigators will contact the Sponsor prior to unblinding any subject's treatment unless in the instance of a medical emergency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sonlicromanol (KH176) (Experimental): Administration of 90 mg sonlicromanol (equivalent to 100 mg sonlicromanol.HCl) twice daily
  Interventions: Drug: Sonlicromanol
- Matching Placebo (Placebo Comparator): Administration of 100 mg matching placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sonlicromanol — Administration of 90 mg sonlicromanol (100 mg sonlicromanol.HCl) twice daily during 52 weeks
  Arms: Sonlicromanol (KH176)
Drug: Placebo — Administration of 100 mg placebo twice daily during 52 weeks
  Arms: Matching Placebo

SUMMARY:
The KHENERFIN study aims to determine whether the study medicine, sonlicromanol, is able to reduce symptoms of fatigue and the impact of fatigue on daily life, and whether sonlicromanol is able to improve physical abilities of people like balance control and lower limb skeletal muscle strength in people with mitochondrial disease.

In this study, the effects of sonlicromanol are compared against a placebo, a tablet identical in appearance and taste but without the active drug. Participants take either sonlicromanol or placebo twice daily for a treatment duration of 52 weeks.

In addition to these primary objectives, the study evaluates the efficacy of sonlicromanol on secondary and exploratory outcomes, as well as its safety and tolerability after one year of treatment.

DETAILED DESCRIPTION:
The KHENERFIN study is investigating the medicine sonlicromanol. The study aims to see if sonlicromanol can reduce symptoms of fatigue and reduce the impact of fatigue on daily life. The study also investigates if sonlicromanol improves physical abilities like balance control and lower limb skeletal muscle strength in people with mitochondrial disease. In addition to these primary objectives, the study evaluates the efficacy of sonlicromanol on selected secondary and exploratory outcomes. It also assesses the safety and tolerability of sonlicromanol.

This study is a placebo controlled, double blind study; the effects of sonlicromanol will be compared with a placebo (study medication that looks like the actual study medicine but contains no active medicine). Neither the participants nor the study team know who is receiving the study medicine or placebo. Participants cannot change their assigned rreatment.

During the screening period, which lasts a maximum of 4 weeks, it is assessed whether the potential participant meets all requirements to participate in the study. Patients who complete the screening phase and are enrolled in the study are randomly (by chance) assigned to receive either the study medicine sonlicromanol or placebo (no active medication). Participants have an equal chance of receiving either sonlicromanol or a placebo. A final follow-up visit is scheduled 2 weeks after taking the last dose of study medication. Total study duration is approximately 60 weeks.

Sonlicromanol will be supplied in tablet form, containing 90 mg of sonlicromanol (equivalent to 100 mg of sonlicromanol.HCl), with the tablets embossed accordingly or provided as a placebo. The study medication must be taken twice daily during the treatment period of 52 weeks. Up to 220 subjects with a confirmed mitochondrial DNA tRNALeu(UUR) 3243A>G mutation will be randomly assigned in a 1:1 ratio to receive either sonlicromanol or placebo.

ELIGIBILITY:
Inclusion criteria

1. Signed Informed Consent
2. Males and females aged ≥18 years with a multi-system primary mitochondrial disease.
3. A confirmed mitochondrial DNA tRNALeu(UUR) m.3243A>G mutation (m.3243A>G PMD) plus an age adjusted heteroplasmy percentage ≥ 20% in white blood cells [=blood heteroplasmy/0.977(age+12)]. Or in urine (urinary epithelial cells), or buccal smear or skeletal muscle (results (obtained per local guidance) ≥ 20% must be available prior to the subject being randomized).
4. Presence of chronic fatigue (not attributable to other etiologies than PMD):

   1. Patient self-reported chronic fatigue for at least 3 months prior to the Screening Visit and recorded in the clinical patient files; AND
   2. Presence of fatigue (raw total score >22), assessed by Neuro-QoL SFv1-F at Screening.
5. Presence of mitochondrial myopathy defined as:

5xSST at Screening and Baseline should be ≥ 11 seconds and participant must demonstrate the ability to complete the test at baseline (i.e., complete the test within 30 seconds).

6. Other Inclusion criteria per protocol.

Exclusion criteria

1. Treatment with any IMP within 3 months (or 5 times the half-life of the IMP, whichever is longer) prior to screening or plans to use an IMP (other than the study intervention) during the study.
2. Bone deformities, motor abnormalities or chronic ulcers that in the opinion of the PI may interfere with and/or confound the interpretation of the subject's performance during the 5 times sit to stand test (5XSST).
3. Surgery of gastrointestinal tract that might interfere with drug absorption. Or severe GI dysmotility, chronic vomiting, diarrhea, bouts of pseudo-obstruction which will impair appropriate IMP absorption in the opinion of the investigator.
4. Clinically significant respiratory disease and/or cardiac disease (medical history or current clinical findings) in the opinion of the investigator.
5. Prior interventional cardiac procedure (e.g., cardiac catheterization, angioplasty/percutaneous coronary intervention, balloon valvuloplasty, etc.) within 3 months prior to screening.
6. QTcF > 450 msec (men) or QTcF > 470 msec (women).
7. Structural heart disease based on cardiac MRI or Echocardiography (e.g., clinically significant valve disease; i.e., aortic or mitral valve stenosis or regurgitation) and/or abnormal conduction (QRS >120 msec, PR > 120 msec), and/or repolarization (QTcF > 450 msec (men) or QTcF > 470 msec (women)). Myocardial function (LVEF <52% in men and < 54% in women), symptomatic ischemic heart disease (inducible ischemia or coronary obstruction), and/or pathologic hypertrophy (e.g. > 15mm septal or posterior wall thickness), that is not well controlled under current specialized care. Subjects with congestive heart failure class II and above should also be excluded.
8. Family history of unexplained/uninvestigated syncope or congenital long and short QT syndrome or sudden death (under the age of 60). ECG evidence of acute or recent ischemia, acute or Recent Myocardial Infraction, atrial fibrillation, high grade AV Blocks (Second Degree AV Block Type II or Third-degree AV Block), complete Heart Block or active conduction system abnormalities with the exception of any of the following:

   1. First degree atrioventricular (AV)-block
   2. Second degree AV-block Type 1 (Mobitz Type 1/Wenckebach type)
   3. Right bundle branch block.
9. History of acute heart failure (within the last 3 months).
10. Higher degree of AV-blocks (AVB II° or III°).
11. Other exclusion criteria per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Neuro-QoL Fatigue Short Form v1 | Screening, Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  Change from baseline compared to placebo at week 52 and at other relevant study visits of the Quality of Life in Neurological Disorders Fatigue Short Form version 1 (Neuro-QoL Fatigue - SF v1): The Neuro-QoL Fatigue SF v1 is an 8-item self-assessment questionnaire evaluating the perception of fatigue and its impact in daily life activities. Each question is scored as following: 1=Never, 2=Rarely, 3=Sometimes, 4=Often, and 5=Always. Total raw scores range from 8-40. T-scores are calculated from the short form scoring table provided in the instruments´ manual. T-score distributions rescale raw scores into standardized scores with a mean of 50 and a standard deviation (SD) of 10. Change from baseline: Negative numbers mean less fatigue, better outcome, positive score means more fatigue, worse outcome.
Five Times Sit-To-Stand Test (5XSST) | Screening, Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  Change from Baseline compared to placebo at week 52 and at other relevant study visits of the 5xSST in total time (in seconds) to complete the 5xSTS. The 5xSST scoring is based on the amount of time (to the nearest decimal in seconds a subject is able to transfer from a seated to a standing position and back to sitting five times. Inability to complete five repetitions without assistance or use of upper extremity support indicates 'failure to perform of test, any modifications should be documented. Participant is directed to stand up straight as quickly as possible 5 times, without stopping in between, keeping arms folded across the chest. When 5xSST is not reached within 30.0 seconds the test is stopped and the actual number of sit to stands reached within those 30 seconds is recorded. Faster times (in sec) denotes better performance.

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) | Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  Change from Baseline at week 52 and at other relevant study visits of the 36-item Short Form Survey Instrument (SF-36). SF36 is a 36-item multidimensional self-report health related quality of life (HRQoL) questionnaire, containing 36 items measuring eight dimensions of HRQoL: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. To score the SF-36, scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100. Standard scoring algorithms yield two distinct, higher-order summary scores: Physical Component Summary (PCS) and Mental Component Summary (MCS). Higher scores on all subscales represent better health and functioning.
The PROMIS Fatigue Primary Mitochondrial Disease Short Form (PROMIS) Fatigue PMD SF) | Screening, Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  Change from baseline at week 52 and at other relevant study visits of the Patient-Reported Outcomes Measurement Information System (PROMIS®) Fatigue Primary Mitochondrial Disease Short Form (PROMIS Fatigue PMD SF). The PROMIS Fatigue Primary Mitochondrial Disease Short Form is a nine-item self-report inventory to assess fatigue symptoms and impacts on daily living measured in PMD. The PROMIS Fatigue PMD SF asks the respondent to rate the experience and impact of fatigue symptoms by asking how often they feel or experienced specific fatigue symptoms in the past seven days on a 5-point rating scale scored as: "never" (1), "rarely" (2), "sometimes" (3), "often" (4), "always" (5). Higher scores indicate greater fatigue severity.
Beck Depression Inventory-2 (BDI-2) | Screening, Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  Change from Baseline compared to placebo at week 52 and at other relevant study visits of the Beck Depression Inventory (BDI). The Beck Depression Inventory (BDI) is a 21-question multiple-choice self-report inventory, for measuring the severity of depression. It is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex. Each answer is scored on a scale value of 0 to 3; higher scores indicate more severe depressive symptoms.
Patient-scored Global Impression of Severity scale (PGI-S) | Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  Change from Baseline compared to placebo at week 52 and at other relevant study visits of the Patient Global Impression of Severity (PGI-S).The Patient scored Global Impression - Severity questionnaire assesses patient's impression of disease severity. The PGI-S item asks the respondent to rate the severity of their PMD symptoms at the time of assessment ("Please choose the response that best describes the severity of your Primary Mitochondrial Disease (PMD) symptoms today") on a 7-point scale scored as: "none" (1), "very mild" (2), "mild" (3), "moderate" (4), "moderately severe" (5), "severe", (6), or "extremely severe" (7). Higher scores indicate a higher level of severity.
Clinician-scored Global Impression of Severity (CGI-S) | Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  Change from Baseline compared to placebo at week 52 and at other relevant study visits of the Clinician Global Impression of Severity (CGI-S). The Clinician scored Global Impression - Severity (CGI-S) scale is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The CGI-S asks the clinician one question: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" which is rated on the following seven-point scale: "normal, not at all ill" (1), "borderline" (2), "mild" (3), "moderate" (4), or "marked" (5), "severe" (6), and "among the most extremely affected patients" (7). This rating is based upon observed and reported symptoms, behaviour, and function at the time of the assessment.Higher scores indicate a higher level of severity.

OTHER OUTCOMES:
Newcastle Mitochondrial Disease Adult Scale (NMDAS) | Baseline (Day 1), Weeks 26, 52 (End of Trial Visit)
  Change from Baseline compared to placebo at week 52 and at other relevant study visits of the Newcastle Mitochondrial Disease Scale for Adults (NMDAS). The NMDAS is a semi-quantitative clinical rating scale designed specifically for all forms of mitochondrial disease. The rating scale encompasses all aspects of mitochondrial disease by exploring several domains: current function, system specific involvement, and current clinical assessment. Each question/item in the NMDAS has a possible score from 0-5. Each of the three section scores are calculated by simply summing the scores obtained for each question in that section, with the higher the score the more severe the disease. Thus, scores can range from 0 to 50 for Sections I and III, and from 0 to 45 for Section II, and from 0 to 145 for Sections I through III. Higher scores indicate a higher level of disease severity.
Brief Pain Inventory Short Form (BPI-SF) | Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  Change from Baseline compared to placebo at week 52 and at other relevant study visits of the Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF is a validated (33) self-administered questionnaire to assess the severity of pain and the impact of pain on the patient's daily functions. BPI-SF evaluates pain severity at its worst, least, and average during the last 24 hours, as well as current pain level, with 0 representing no pain and 10 the worst pain imaginable. Seven items measuring interference with daily functioning (general activity, walking, work, mood, relations with others, sleep, and enjoyment of life) are also assessed on an 11-point scale, where 0 represents no interference and 10 complete interferences. The scores can be averaged to the two components of the BPI SF score, the Pain Severity Index and the Pain Interference Index. Higher scores indicate a higher level of severity and impact of pain.
Health Economics and Outcomes Research (HEOR) Assessments: EQ-5D-5L | Screening, Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit) and at week 54 (Follow-up)
  Change from Baseline compared to placebo at week 52 and at other relevant study visits of the EQ-5Dimension-5 Level (EQ-5D-5L). The EQ-5D-5L is a self-report health-related quality of life (HRQoL) instrument consisting a descriptive system and a visual analogue scale (EQ-VAS). The descriptive system that defines health in five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response categories (levels): no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ-VAS records the respondent's self-rated health on a vertical VAS. The respondents can report their perceived health status with a grade ranging from 0 ('the worst health you can imagine') to 100 ('the best health you can imagine'). A higher score denotes a worse health state.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Screening, Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  Change from Baseline compared to placebo at week 52 and at other relevant study visits of the Columbia-Suicide Severity Rating Scale (C-SSRS). The instrument assesses severity of suicidal ideation ("severity subscale"), rated on a 5-point ordinal scale, the intensity of ideation subscale ("intensity subscale"), comprising 5 items, rated on a 5-point ordinal scale: frequency, duration, controllability, deterrents, and reason for ideation, resulting in 0-25 score range summed from five items, with higher scores indicating more severe suicidal ideation. A score of 0 indicates that no suicide ideation is present. The behaviour subscale is a nominal scale including actual, aborted, and interrupted attempts; preparatory behaviour; and self-injurious behaviour. The lethality subscale assesses actual attempts; actual lethality rated on a 6-point ordinal scale. Higher scores indicate a higher level of severity.
Gastro-Intestinal symptoms. | Through week 52
  Change from Baseline compared to placebo on the number of gastro-intestinal complaints, intensity and duration. The number of gastro-intestinal complaints/month will be captured, starting at screening until (and including) the week 52 visit. For this purpose the Gastro-Intestinal symptoms questionnaire will be used.
Seizure episodes | Through week 52
  Change from Baseline compared to placebo on the number of seizures, intensity and duration and on the use of medication. Seizure data (e.g., occurrence, duration, intensity severity; and any use of migraine medication) are captured daily through a daily headache-diary.
Safety and tolerability assessed by nature, frequency and severity of treatment emergent adverse events (TEAEs) | Through Week 52
  Safety and tolerability assessed by nature, frequency and severity of treatment emergent adverse events (TEAEs) Treatment emergent adverse events will be coded using medical dictionary for regulatory activities (MedDRA). A TEAE is defined as an adverse event (AE) observed after starting administration of the investigational product (IP) to 14 days after last dose of IP. An AE is any untoward medical occurrence in a participant, temporally associated with the use of IP, whether or not considered related to the IP. An AE can therefore be any unfavourable and unintended, symptom, or disease (new or exacerbated) temporally associated with the use of IP.
Safety: 12 lead ECG parameters: QRS duration (milliseconds) | Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  12 lead ECG parameter data QRS duration (milliseconds) will be summarised.
Safety: 12 lead ECG parameters: QRS morphology (peak, axis) | Baseline (Day 1), Weeks 13, 26, 39, 52 (End of Trial Visit)
  12 lead ECG parameter data QRS morphology (peak, axis) will be summarised.
Safety: 12 lead ECG parameters: QTcF (Fridericia) | Screening, Baseline (Day 1), Day 6, Weeks 4, 8, 13, 26, 39, 52 (End of Trial Visit), 54 (Safety FU)
  12 lead ECG parameter data QTcF (Fridericia) will be summarised.
Safety: 12 lead ECG parameters: PQ interval: milliseconds (ms)) | Screening, Baseline (Day 1), Day 6, Weeks 4, 8, 13, 26, 39, 52 (End of Trial Visit), 54 (Safety FU)
  12 lead ECG parameter data PQ intervals (milliseconds) will be summarised.
Safety: 12 lead ECG parameters: Heart rate: beats per minute (bpm) | Screening, Baseline (Day 1), Day 6, Weeks 4, 8, 13, 26, 39, 52 (End of Trial Visit), 54 (Safety FU)
  12 lead ECG parameter data Heart rate (beats per minute (bpm) be summarised.
Safety: 12 lead ECG parameters: Tpeak-Tend interval | Screening, Baseline (Day 1), Day 6, Weeks 4, 8, 13, 26, 39, 52 (End of Trial Visit), 54 (Safety FU)
  12 lead ECG parameter data (Tpeak-Tend interval) will be summarised.
Safety: 12 lead ECG parameters: T wave morphology (peak, symmetry) | Screening, Baseline (Day 1), Day 6, Weeks 4, 8, 13, 26, 39, 52 (End of Trial Visit), 54 (Safety FU)
  12 lead ECG parameter data T-wave morphology (symmetry) will be summarised.
Safety: Incidence of laboratory abnormalities, based on haematology, clinical chemistry, and urinalysis test results | Screening, Baseline (Day 1), Weeks 4, 8, 13, 26, 39, 52 (End of Trial Visit)
  Incidence of laboratory abnormalities outside the clinical reference ranges based on haematology, serum biochemistry, and urinalysis test
Safety: Vital signs abnormalities and/or AEs | Screening, Baseline (Day 1), Weeks 26, 52 (End of Trial Visit),54 (Safety FU)
  Incidence of clinically significant vital sign values.
Pharmacokinetics: Tmax (hours) | Week 39: pre-dose, and at 1, 2, 4, 6, 8 hours post dosing.
  Tmax: Time to reach maximum (peak) plasma concentration following drug administration (hours)
Pharmacokinetics: Cmax (ng/mL) | Week 39: pre-dose, and at 1, 2, 4, 6, 8 hours post dosing.
  Maximum (peak) plasma drug concentration in ng/mL
Pharmacokinetics: Ctrough (ng/mL) | Week 39: pre-dose, and at 1, 2, 4, 6, 8 hours post dosing.
  Plasma concentration (measured concentration at the end of a dosing interval at steady state in ng/mL
Pharmacokinetics: AUCinf (h*ng/mL) | Week 39: pre-dose, and at 1, 2, 4, 6, 8 hours post dosing.
  Area under the plasma concentration time curve from time zero to infinity in h*ng/mL
Pharmacokinetics: AUCtau (h*ng/mL) | Week 39: pre-dose, and at 1, 2, 4, 6, 8 hours post dosing.
  Area under the plasma concentration time curve in h*ng/mL
Pharmacokinetics: T1/2 (hours) | Week 39: pre-dose, and at 1, 2, 4, 6, 8 hours post dosing.
  Terminal Elimination Half-life

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cleveland Clinic Neurological Institute Mellen Center, Cleveland, Ohio
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Rigshospitalet, University of Copenhagen, Kopenhagen, Region Sjælland, Denmark
- France (2):
  - CHU de Bordeaux - Hôpital Pellegrin Service Gynecologie Obstetrique, Bordeaux, Gironde
  - Groupe Hospitalier Pitie-Salpetriere - Charles-Foix Clinical Investigation Center Paris-Est, Paris, Paris
- Klinikum der Universität München Friedrich-Baur-Institut, München, Germany
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Milano, Italy
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands
- University College London Hospitals NHS Foundation Trust National Hospital for Neurology and Neurosurgery, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided